CLINICAL TRIAL: NCT04590573
Title: The Effects of Cognitive-behaviour Couple Therapy and Emotionally Focused Couple Therapy for Chinese Couples With a Depressed Partner in Hong Kong: A Comparison to a Social Activity Control Group
Brief Title: Cognitive Behavioural Couple Intervention Therapy for Chinese Couples With a Depressed Partner
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Chinese University of Hong Kong (Other); City University of Hong Kong (Other); York University (Other)
Responsible Party: Principal Investigator, Professor Daniel Fu-Keung Wong, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBCT
Record Dates: First submitted 2020-10-04; First posted 2020-10-19 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBCT (Experimental): Cognitive behavioural couple therapy (CBCT), 5-session
  Interventions: Behavioral: Cognitive behavioural couple therapy (CBCT), Emotion focused couple therapy (EFCT), Wait-list control (Control)
- EFCT (Experimental): Emotion focused couple therapy (EFCT), 5-session
  Interventions: Behavioral: Cognitive behavioural couple therapy (CBCT), Emotion focused couple therapy (EFCT), Wait-list control (Control)
- Control (Active Comparator): Social activity wait-list groups (Control), 5-session
  Interventions: Behavioral: Cognitive behavioural couple therapy (CBCT), Emotion focused couple therapy (EFCT), Wait-list control (Control)

INTERVENTIONS:
Behavioral: Cognitive behavioural couple therapy (CBCT), Emotion focused couple therapy (EFCT), Wait-list control (Control) — 5 sessions in CBCT, EFCT and Control (3 hours per session), 6-8 pairs of couples per group and around 7 groups will be held.

SUMMARY:
Understanding depression from a relational perspective maybe more meaningful in Chinese culture due to the different values and beliefs among Chinese comparing to those of the Western cultures. The PI and his associates developed a Cognitive Behavioural Couple Therapy model for Chinese couples with a depressed partner receiving mental health services in a community mental health centre in Hong Kong between 2018 and 2019. With consideration of the limitations in a pilot study conducted by the PI, modifications are made in the current study. This study aims to evaluate the effectiveness of a cognitive behavioural couple therapy model for Chinese couples with a depressed partner in Hong Kong. A comparison approach involving cognitive behavioural couple therapy (CBCT), emotional focused couple therapy (EFCT) and a wait-list control group on their short-term and long-term effects, as well as differential benefits will be examined.

A set of questionnaires will be filled out by the 135 participants (45 in each arm) before the intervention (T0), after the intervention (T1), and 6-month after the intervention (T2). It is hypothesized that comparing to the control group, participants in CBCT and EFCT conditions will have greater improvements in outcomes at T1 and T2. There will be differential therapeutic effects of CBCT and EFCT on the various outcomes. Different mediating effects behind the changes in the outcomes in the two conditions will be examined.

The study will contribute to the current literature by evaluating the effectiveness of culturally-attuned CBCT and EFCT. New insights will be added to the current therapeutic approaches for couples with a depressed partner.

A sets of questionnaires will be assessed before the intervention (T0), after the intervention (T1), and 6-month after the intervention (T2). It is hypothesized that comparing to the control group, participants in CBCT and EFCT conditions will have greater improvements in outcomes at T1 and T2. Also, they may receive differential therapeutic effects of CBCT and EFCT on different outcomes. Different mediating effects behind the changes in the outcomes will be examined.

The study will contribute to the current literature by evaluating the effectiveness of culturally-attuned CBCT and EFCT. Insights may be provide to the current therapeutic approach for couples with depressed partners.

ELIGIBILITY:
Inclusion Criteria:

* Chinese couples aged 18 to 65
* Able to understand Cantonese or Chinese
* One of the couples having a diagnosis of DSM-V Major Depressive Disorder (MDD)

Exclusion Criteria:

* Neurological disease or damage that would compromise cognitive functioning
* Suicidal attempts or ideation in the past 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Patient Health Questionnaire-9 at 2 months (post-intervention) and 8 months (6 months after intervention) | Day 0 (Baseline), Month 2 (Post-intervention), Month 8 (6-month follow-up)
  To assess frequency of depressive symptoms of the participants during the preceding 2 weeks. The 9 items are rated on a 3-point scale from 0 (not at all) to 3 (nearly every day). The range of the scale is 0 to 27. Higher scores indicated more depressive symptoms.
Change from Baseline Depression Anxiety Stress Scales-Chinese Version at 2 months (post-intervention) and 8 months (6 months after intervention) | Day 0 (Baseline), Month 2 (Post-intervention), Month 8 (6-month follow-up)
  To assess the emotional states of depression, anxiety and stress in the participants. The 21 items are rated on a 4-point scale from 0 (not applicable) to 3 (very applicable). Sum scores are computed by adding up the scores of each item and then multiplying by 2. The range of the scale is from 0 to 120. Higher scores indicated higher levels of depression, anxiety and stress.

SECONDARY OUTCOMES:
Change from Baseline Dyadic Adjustment Scale at 2 months (post-intervention) and 8 months (6 months after intervention) | Day 0 (Baseline), Month 2 (Post-intervention), Month 8 (6-month follow-up)
  To evaluate 4 dimensions of marital quality of the participants (Consensus, Cohesion, Satisfaction and Affectional Expression). The range of the scale is 0 to 151. Lower total scores indicate greater distress in marital relationships.
  The 15 items of Consensus are rated on a 6-point scale from 0 (totally agree) to 5 (totally disagree). Two of the 6 items of Cohesion are rated on a 5-point scale from 0 (daily/all) to 4 (never) while the remaining 4 items on a 6-point scale from 0 (never) to 5 (always). Seven of the 9 items of Satisfaction are rated on a 6-point scale from 0 (anytime) to 5 (never) while one of the remaining items asked the participants to describe their marriage from 7 choices from "extremely unhappy" to "perfect". The last item included 6 sentences about views on the marital relationships and the participants are asked to choose the best one describing their thoughts. The 2 items of Affectional Expression are answered by "yes" or "no".
Change from Baseline Marital Satisfaction with Life Scale at 2 months (post-intervention) and 8 months (6 months after intervention) | Day 0 (Baseline), Month 2 (Post-intervention), Month 8 (6-month follow-up)
  To measure the subjective evaluation of one's satisfaction in life. The 5 items are rated on a 7-point scale from 1(strongly disagree) to 7(strongly agree). The range of the scale is 5 to 35. Higher scores represent greater life satisfaction.
Change from Baseline Difficulties in Emotion Regulation Scale-Short Form at 2 months (post-intervention) and 8 months (6 months after intervention) | Day 0 (Baseline), Month 2 (Post-intervention), Month 8 (6-month follow-up)
  To assess individuals' emotion dysregulation patterns. The 18 items are rated on a 5-point scale from 1 (almost never) to 5 (almost always). The range of the scale is 18 to 90. Higher scores indicate greater emotion dysregulation.
Change from Baseline Relationship Belief Inventory at 2 months (post-intervention) and 8 months (6 months after intervention) | Day 0 (Baseline), Month 2 (Post-intervention), Month 8 (6-month follow-up)
  To measure unrealistic beliefs about marriage of the participants. The 40 items are rated on 6-point scale from 0 (strongly believe the statement is false) to 5 (strongly believe the statement is true). The range of the scale is 0 to 200. Higher scores indicate a greater adherence to the related beliefs in marriage.

CONTACTS AND LOCATIONS:
Overall Officials: Fu Keung Daniel Wong, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
There is a platform for data sharing in the university
Time Frame: after the research project is completed
Access Criteria: based on the policy of the university
URL: https://libguides.lib.hku.hk/researchdata/datahub